

# HOJA DE INFORMACIÓN AL PACIENTE ADULTO

Versión: 1 Fecha de la versión: 28 de noviembre de 2022

Investigador/a Principal: Antonio J Conde Moreno. Servicio de Oncología Radioterápica. 649039866. antoniojconde@gmail.com

CENTRO: Hospital Universitario y Politécnico la Fe

Título del proyecto de investigación: Desarrollo de una crema protectora frente a

las radiodermitis causadas por la radioterapia.

ACRÓNIMO: RADIOCREMVAL

#### 1. INTRODUCCIÓN:

Nos dirigimos a usted para informarle sobre un estudio en el que se le invita a participar. El estudio ha sido aprobado por el Comité de Ética de la Investigación con medicamentos del Hospital Universitario y Politécnico La Fe (CEIm La Fe).

Nuestra intención es tan sólo que usted reciba la información correcta y suficiente para que pueda evaluar y juzgar si quiere o no participar en este estudio. Para ello lea esta hoja informativa con atención y nosotros le aclararemos las dudas que le puedan surgir después de la explicación. Además, puede consultar con las personas que considere oportunas.

# 2. PARTICIPACIÓN VOLUNTARIA:

Debe saber que su participación en este estudio es voluntaria y que puede decidir no participar y retirar el consentimiento en cualquier momento, sin que por ello se altere la relación con su médico ni se produzca perjuicio alguno en su tratamiento.

# 3. DESCRIPCIÓN GENERAL DEL ESTUDIO:

El estudio consiste en ensayo de una crema radioprotectora y radiomitigadora para la reducción de la radiodermitis en piel, en pacientes sometidos a tratamiento de radioterapia externa de carcinoma de células escamosas de tumores de cabeza y cuello (SCCHN).

El objetivo principal de nuestra formulación es obtener una reducción (en la progresión a radiodermitis grado 3-4) en pacientes que sufren dermatitis aguda por radiación de grado 3 o 4 a grado 2, evaluada el último día de tratamiento. Retraso en aparición de radiodermitis grado 2 respecto al grupo placebo así como disminución de esta en más de un 10%. Además de este objetivo principal, en este proyecto hay una serie de objetivos secundarios, como la comparación del porcentaje de pacientes con radiodermitis, el grado de toxicidad y el porcentaje de casos con radiodermitis grado 2 o superior en los pacientes sometidos a los diferentes tratamientos, en la muestra total y estratificada por número de sesiones de radioterapia al mes y al finalizar el



tratamiento. También queremos evaluar y comparar el tiempo para la aparición de cada grado de reacción cutánea; identificar la frecuencia y localización de las características específicas de las radiodermitis. Otro objetivo secundario es la calidad de vida relacionada con la salud percibida por los pacientes al inicio y al término de la radioterapia. Evaluar y comparar los síntomas locales descritos por los pacientes durante el tratamiento radioterápico. Por último, se quiere verificar y comparar la temperatura de la zona irradiada mediante un termógrafo, en las 4 visitas que realizará el paciente.

La metodología va a consistir en la distribución de los pacientes en dos grupos, todos los pacientes llevan tratamiento para la radiodermitis. Los paciente son clasificados aleatoriamente en estos grupos. A un grupo de pacientes se les aplicará la crema standard of care y al otro grupo la crema de estudio experimental. Esta crema de estudio está clasificada por la AEMS como cosmecéutico, es decir, la finalidad de esta crema es mantener las condiciones de la piel en buen estado. Las cremas en los dos grupos se aplicarán 2 días antes y durante la radioterapia, 2 veces al día, hasta el final del tratamiento. Los pacientes realizarán 4 visitas al servicio de oncología radioterápica, a los 7 días, a las 3-4 semanas, al finalizar el tratamiento y 2 semanas después del tratamiento. Previamente a estas sesiones, donde se valorarán una serie de parámetros clínicos de rutina en este servicio, habrá una primera visita donde se explicará al paciente el proyecto de investigación, se le entregará la hoja de información y el consentimiento informado.

En las revisiones periódicas a los pacientes, además de la valoración de la radiodermitis con la escala clínica CTCAE del Instituto Nacional del Cáncer clasificación (V.4.03).8-10, y como novedad en este proyecto, se realizarán las encuestas de calidad en relación a la toxicidad por radiodermitis y la valoración objetiva de la temperatura de la piel mediante un termógrafo.

Los sujetos pueden retirar su consentimiento como se indica en esta hoja de información en cualquier momento y sin perjuicio. Adicionalmente, el investigador puede retirar a un sujeto si, según la opinión clínica del investigador, está en el mejor interés del sujeto o si el sujeto no puede cumplir con los requisitos del protocolo. En relación a los inconvenientes y riesgos derivados del estudio, hay una serie de motivos para detener el estudio, y uno de ellos es si la incidencia de la radiodermitis es inaceptable, no esperable. Es decir, caso de que el paciente presente radiodermatitis de grado 1 o 2, el protocolo del estudio se mantendrá inalterado con la continuación de la aplicación de la crema, ya que el tratamiento estándar de estas lesiones es la aplicación de hidratantes tópicos, función ya desempeñada por la crema estudiada. En caso de que el paciente presente radiodermatitis de grado 3 o 4, la radioterapia y la aplicación de la crema podrán ser suspendidas por el radioterapeuta hasta que la lesión de piel mejore; el tratamiento tópico de las lesiones corresponderá a sus características, conforme con el protocolo institucional. El paciente deberá continuar aplicando la crema en las regiones irradiadas no afectadas por la lesión.

El número total de sujetos que se incluirá en el estudio es de 82.

Las responsabilidades del sujeto que participe en el estudio, le serán explicadas el primer día de visita clínica, con la entrega de esta hoja de información y la firma del consentimiento. El paciente se debe comprometer a aplicarse las cremas, en los tiempos y las pautas indicadas por los investigadores. Además, se deben comprometer a notificar cualquier evento adverso que le suceda o cualquier cambio en su medicación.



# 4. BENEFICIOS Y RIESGOS DERIVADOS DE SU PARTICIPACIÓN EN EL ESTUDIO:

La dermatitis radioinducida es uno de los efectos secundarios más frecuentes de la radioterapia.

Se considera RADIODERMITIS al conjunto de lesiones cutáneas que aparecen tras la exposición de la piel a radiaciones ionizantes, bien con fines terapéuticos o de forma accidental. Existen varias escalas para la clasificación de la severidad de las dermitis inducidas por radiación. En la actualidad, no existe un estándar de cuidados ni hay directrices para la prevención y el tratamiento de la dermatitis aguda por radiación. La mayoría de los tratamientos utilizados actualmente son adecuados, pero no óptimos en lo que respecta a eficacia y seguridad/tolerancia. Además, la evidencia clínica que respalda su uso es limitada.

A los pacientes se les proveerá de las cremas que se necesitan para el estudio de manera gratuita para todo el tiempo del estudio. Las cremas standard of care son comerciales y de uso habitual para intentar mitigar el efecto de la radioterapia. La crema experimental no está comercializada.

Como beneficio por su participación, la valoración de la radiodermitis se realizará más exhaustivamente, con un mayor control y con equipamiento novedoso que hasta ahora no se utilizaba para valorar estas posibles lesiones en la piel.

Las cremas utilizadas en este estudio no están contraindicadas en el embarazo.

Debe saber que su participación en este estudio puede no aportarle beneficios directos.

# 5. TRATAMIENTOS ALTERNATIVOS:

No existen alternativas terapéuticas para estos pacientes. Las cremas comerciales que se les proporcionan inducen efectos radiomitigadores en la piel afecta en un % muy pequeño (ver arriba).

#### 6. Nº DE URGENCIA PARA PROBLEMAS DEL ESTUDIO:

En caso de que desee formular preguntas acerca del estudio o daños relacionados con el mismo, puede contactar con el médico del estudio, el Dr. Antonio J. Conde, en el número de teléfono 961245108.

# 7. CONFIDENCIALIDAD:

El tratamiento, la comunicación y la cesión de los datos de carácter personal de todos los sujetos participantes se ajustará a lo dispuesto en la Ley Orgánica 3/2018, de 5 de diciembre de protección de datos y garantía de los derechos digitales y en el Reglamento (UE) 2016/679 del Parlamento europeo y del Consejo de 27 de abril de 2016 de Protección de Datos (RGPD). De acuerdo a lo que establece la legislación mencionada, usted puede ejercer los derechos de acceso, modificación, oposición,



cancelación de datos, limitar el tratamiento de datos que sean incorrectos y solicitar una copia o que se trasladen a un tercero (portabilidad) para lo cual deberá dirigirse al investigador/a principal del estudio o al/a la Delegado/a de Protección de Datos de la Institución, con quién podrá comunicarse a través del teléfono y/o dirección de correo electrónico: oncoradi lafe@gya.es y teléfono 961245108.

Le recordamos que los datos no se pueden eliminar, aunque deje de participar en el estudio, para garantizar la validez de la investigación y cumplir con los deberes legales. Así mismo tiene derecho a dirigirse a la Agencia de Protección de Datos si no quedara satisfecho.

Tanto el Centro como el Promotor son responsables respectivamente del tratamiento de sus datos y se comprometen a cumplir con la normativa de protección de datos en vigor. Los datos recogidos para el estudio estarán identificados mediante un código, de manera que no se incluya información que pueda identificarle, y sólo su médico del estudio/colaboradores podrá relacionar dichos datos con usted y con su historia clínica. Por lo tanto, su identidad no será revelada a ninguna otra persona salvo a las autoridades sanitarias, cuando así lo requieran o en casos de urgencia médica. Los Comités de Ética de la Investigación con medicamentos, los representantes de la Autoridad Sanitaria en materia de inspección y el personal autorizado por el Promotor, únicamente podrán acceder para comprobar los datos personales, los procedimientos del estudio clínico y el cumplimiento de las normas de buena práctica clínica (siempre manteniendo la confidencialidad de la información).

El / la Investigador/a y el Promotor están obligados a conservar los datos recogidos para el estudio al menos hasta 25 años tras su finalización. Posteriormente, su información personal solo se conservará por el centro para el cuidado de su salud y por el promotor para otros fines de investigación científica si usted hubiera otorgado su consentimiento para ello, y si así lo permite la ley y requisitos éticos aplicables.

Sólo se tramitarán a terceros y a otros países los datos recogidos para el estudio, que en ningún caso contendrán información que le pueda identificar directamente, como nombre y apellidos, iniciales, dirección, nº de la seguridad social, etc... En el caso de que se produzca esta cesión, será para los mismos fines del estudio descrito y garantizando la confidencialidad como mínimo con el nivel de protección de la legislación vigente en nuestro país.

# 8. COMPENSACIÓN ECONÓMICA:

El promotor del estudio es el responsable de gestionar la financiación del mismo, por lo que su participación en éste no le supondrá ningún gasto.

# 9. OTRA INFORMACIÓN RELEVANTE:

Cualquier nueva información que se descubra durante su participación y que pueda afectar a su disposición para participar en el estudio, le será comunicada por su médico lo antes posible.

Si usted decide retirar el consentimiento para participar en este estudio, no se añadirá ningún dato nuevo a la base de datos y, en caso de que se hubieran recogido



muestras, puede exigir la destrucción de todas las muestras identificables, previamente obtenidas, para evitar la realización de nuevos análisis.

También debe saber que puede ser excluido del estudio si el promotor o los investigadores del mismo lo consideran oportuno, ya sea por motivos de seguridad o porque consideren que usted no está cumpliendo con los procedimientos establecidos. En cualquiera de los casos, usted recibirá una explicación adecuada del motivo por el que se ha decidido su retirada del estudio.

El promotor podrá suspender el estudio siempre y cuando sea por alguno de los supuestos contemplados en la legislación vigente.

Al firmar la hoja de consentimiento adjunta, se compromete a cumplir con los procedimientos del estudio que se le han expuesto. Cuando acabe su participación recibirá el mejor tratamiento disponible y que su médico considere el más adecuado para su enfermedad.



# **CONSENTIMIENTO POR ESCRITO**

Título del estudio: Desarrollo de una crema protectora frente a las radiodermitis causadas por la radioterapia.

| Yo, | (nombre y ap | pellidos). |
|---|---|---|
| <ul> <li>He leído la hoja de información que se me h</li> </ul> | | e se me ha entregado. |
| • | He podido hacer preguntas sobre e | el estudio. |
| • | He recibido suficiente información sobre el estudio.<br>He hablado con: (nombre del Investigador/a) | |
| • | | |
| • | Comprendo que mi participación es | s voluntaria. |
| • | Recibiré una copia firmada y fecha | da de este documento de consentimiento informado. |
| Comp | orendo que puedo retirarme del estud | lio: |
| Comp | 1º Cuando quiera | iio. |
| | 2º Sin tener que dar explicaciones. | |
| | 3º Sin que esto repercuta en mis cu | |
| Presto | o libremente mi conformidad para pa | rticipar en el estudio. |
| Firma | del Participante | Firma del Investigador/a |
| Nombre: | | Nombre: |
| recna | ı:/ | Fecha:// |
| | o que me comuniquen la información<br>mí salud: <b>Sí No</b> | derivada de la investigación que pueda ser relevante |
| Firma del representante | | Fecha:/(Nombre, firma y fecha |
| ae puno | y letra del representante legal) | |
| Firma | del investigador/a: | Fecha:/ |
| | | ación derivada de las pruebas genéticas realizadas<br>e incluyan este tipo de pruebas, siempre que estén |
| | | para la salud del paciente): 🗌 <b>Sí</b> 🦳 <b>No</b> |
| Firma del representante | | Fecha:/(Nombre, firma y fecha |
| de puño | y letra del representante legal) | |
| Firma del investigador/a: | | Fecha:// |